CLINICAL TRIAL: NCT02653313
Title: A Non-controlled, Single Arm, Open Label, Phase II Study of Intravenous and Intratumoral Administration of ParvOryx in Patients With Metastatic, Inoperable Pancreatic Cancer
Brief Title: Parvovirus H-1 (ParvOryx) in Patients With Metastatic Inoperable Pancreatic Cancer
Acronym: ParvOryx02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oryx GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ParvOryx02
Record Dates: First submitted 2015-12-04; First posted 2016-01-12 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Pancreatic Ductal
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ParvOryx (Experimental): ParvOryx given intravenously on four consecutive days (day 1 to 4) and intrametastatic six to thirteen days thereafter (day 7, 10 or 14).
  Interventions: Drug: Parvovirus H-1 (H-1PV)

INTERVENTIONS:
Drug: Parvovirus H-1 (H-1PV) — Parvovirus H-1 administered at three increasing dose levels , according to the following schedule: i) 4 daily intravenous infusions of 10% of the total dose over 2 hours on 4 consecutive days, ii) direct injection of 60% of the total dose into a hepatic metastasis of the pancreatic cancer.
  The total dose levels are: 1E09, 5E09 and 1E10 pfu.
  Other Names: ParvOryx

SUMMARY:
Investigation on safety, tolerability and efficacy of parvovirus H-1 (ParvOryx) in subjects suffering from metastatic, inoperable pancreatic cancer with at least one hepatic metastasis.

DETAILED DESCRIPTION:
Investigation on safety, tolerability and efficacy of parvovirus H-1 (ParvOryx) in subjects suffering from metastatic, inoperable pancreatic cancer with at least one hepatic metastasis.

Initially four equal doses of ParvOryx will be administered intravenously on four consecutive days. Seven to fourteen days after the first intravenous administration the drug will be injected directly in a hepatic metastasis of the pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 year,
2. Ability to give informed consent,
3. Histologically confirmed pancreatic ductal adenocarcinoma (PAD) with at least one measurable hepatic metastasis according to RECIST 1.1,
4. Disease progression despite first line therapy (whatever chemotherapy regimen),
5. Eligibility for second line chemotherapy with gemcitabine,
6. ECOG performance scale 0 or 1,
7. Consent for the sampling and investigations of biological specimens as scheduled by the trial protocol,
8. Adequate bone marrow function: neutrophils >1.5 x 1E09/L, platelets >100 x 1E09/L, hemoglobin >9.0 g/dL,
9. Liver function tests (LFT) within the following range: Bilirubin <3 x ULN (Upper Limit of Normal); ASAT and ALAT <5 x ULN,
10. Adequate renal function: Creatinine <1.5 g/dL,
11. Adequate blood clotting: aPTT <39 sec, INR <1.2,
12. Normal thyroid function, i.e. TSH, fT3 and fT4 within the normal range (TSH: 0.4 - 4.0 mU/l, fT3: 2.0 - 4.2 ng/l, fT4: 8 - 18 ng/l)
13. Negative serology for HIV, HBV and HCV,
14. Negative Beta-HCG test in blood in woman of childbearing potential,
15. Use of adequate contraception in both genders, i.e. use of double-effective method of contraception for the entire participation in the trial.

Exclusion Criteria:

1. Eligibility for surgical treatment,
2. Symptomatic cerebral, pulmonal, and/or osseous metastases,
3. Peritoneal carcinosis,
4. Liver cirrhosis,
5. Splenectomy,
6. Relevant respiratory impairment, corresponding to the grade IV or V of the MRC Breathlessness Scale (stops for breath after walking about 100 meters or after a few minutes on level ground, or too breathless to leave the house, or breathless when undressing),
7. Positive anti-drug antibodies (ADAs) against ParvOryx,
8. Hospitalization due to other conditions than the pancreatic cancer within the last 3 months,
9. Chemotherapy within 2 weeks prior to the first administration of the IMP,
10. Signs of active, systemic infection within 7 days prior to the study inclusion (clinical symptoms (cough, running nose, burning sensation while urinating, apparent skin or wound infection) and/or increase of fever and/or deterioration of infection-specific laboratory parameters beyond changes apparently driven by the underlying pancreatic cancer),
11. Radiotherapy within 6 weeks prior to the study inclusion,
12. Contraindications for CT,
13. Known allergy to iodinated contrast media,
14. Participation in another interventional trial within the last 30 days,
15. Presumed contact with pregnant women and/or infants <12 months of age within two months after the first administration of the IMP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-12; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the IMP | Up to 6 months after treatment beginning
  Parameter: findings in physical examinations
Safety and tolerability of the IMP | Up to 6 months after treatment beginning
  Parameters: chosen laboratory parameters
Safety and tolerability of the IMP | Up to 6 months after treatment beginning
  Parameter: ECG
Safety and tolerability of the IMP | Up to 6 months after treatment beginning
  Parameter: adverse events
Humoral immuneresponse to the IMP | Up to 6 months after treatment beginning
  Parameter: Serum concentration of anti-drug antibodies (ADA)
Pharmacokinetics of viral genomes [Vg] | Up to 6 months after treatment beginning
  Parameter: Cmax in blood
Pharmacokinetics of viral genomes [Vg] | Up to 6 months after treatment beginning
  Parameter: AUC in blood
Shedding of viral genomes [Vg] | Up to 6 months after treatment beginning
  Parameter: Concentration of Vg in feaces
Shedding of viral genomes [Vg] | Up to 6 months after treatment beginning
  Parameter: Concentration of Vg in urine
Shedding of viral genomes [Vg] | Up to 6 months after treatment beginning
  Parameter: Concentration of Vg in saliva

SECONDARY OUTCOMES:
Histo-immuno-pathological effects of the IMP in the hepatic metastasis | Up to 2 months after treatment beginning
  Parameter: extent of tumor necrosis
Histo-immuno-pathological effects of the IMP in the hepatic metastasis | Up to 2 months after treatment beginning
  Parameter: density of tumor infiltrating cells
Histo-immuno-pathological effects of the IMP in the hepatic metastasis | Up to 2 months after treatment beginning
  Parameter: tissue content of cytokines
Histo-immuno-pathological effects of the IMP in the hepatic metastasis | Up to 2 months after treatment beginning
  Parameter: tissue content of chemokines
Extent of virus replication in the hepatic metastasis | Up to 2 months after treatment beginning
  Parameters: quantification of NS-1 protein in the metastatic tissue
Cellular immune response against viral proteins | Up to 6 months after treatment beginning
  Parameter: ELISPOT
Cellular immune response against viral proteins | Up to 6 months after treatment beginning
  Parameter: FACS
Clinical outcome | Up to 6 months after treatment beginning
  Parameters: PFS, OS
Clinical outcome | Up to 6 months after treatment beginning
  Parameter: Serum concentration of CA19-9

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Huber, Dr., Study Director — Oryx GmbH & Co. KG; Guy Ungerechts, Prof. Dr. Dr., Principal Investigator — National Center for Tumor Diseases, Heidelberg
Locations (1):
- National Center for Tumor Diseases (NCT), Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Hajda J, Lehmann M, Krebs O, Kieser M, Geletneky K, Jager D, Dahm M, Huber B, Schoning T, Sedlaczek O, Stenzinger A, Halama N, Daniel V, Leuchs B, Angelova A, Rommelaere J, Engeland CE, Springfeld C, Ungerechts G. A non-controlled, single arm, open label, phase II study of intravenous and intratumoral administration of ParvOryx in patients with metastatic, inoperable pancreatic cancer: ParvOryx02 protocol. BMC Cancer. 2017 Aug 29;17(1):576. doi: 10.1186/s12885-017-3604-y. PMID 28851316
- [Background] Hajda J, Leuchs B, Angelova AL, Frehtman V, Rommelaere J, Mertens M, Pilz M, Kieser M, Krebs O, Dahm M, Huber B, Engeland CE, Mavratzas A, Hohmann N, Schreiber J, Jager D, Halama N, Sedlaczek O, Gaida MM, Daniel V, Springfeld C, Ungerechts G. Phase 2 Trial of Oncolytic H-1 Parvovirus Therapy Shows Safety and Signs of Immune System Activation in Patients With Metastatic Pancreatic Ductal Adenocarcinoma. Clin Cancer Res. 2021 Oct 15;27(20):5546-5556. doi: 10.1158/1078-0432.CCR-21-1020. Epub 2021 Aug 23. PMID 34426438